CLINICAL TRIAL: NCT04968639
Title: The Characteristic of Axial Pain After Open-door Laminoplasty in Patients With Degenerative Cervical Spine Myelopathy and the Correlation With EEG Analysis: a Prospective Cohort Study.
Brief Title: The Characteristic of Axial Pain and EEG Analysis of Patients After Laminoplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019197
Record Dates: First submitted 2021-06-27; First posted 2021-07-20 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Cervical Myelopathy
Keywords: Cervical Myelopathy; Axial Pain; Electroencephalogram Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Axial pain positive group: Postoperative VAS score ≥ 3 points at 3-month follow-up
- Axial pain negative group: Postoperative VAS score ≤ 2 points at 3-month follow-up

SUMMARY:
The characteristic of axial pain and EEG analysis of patients after laminoplasty

DETAILED DESCRIPTION:
The characteristic of axial pain after open-door laminoplasty in patients with degenerative cervical spine myelopathy and the correlation with electroencephalogram analysis: a prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18~70 years.
* Diagnosed as degenerative cervical spine myelopathy.
* Must receive C3-C7 open-door laminoplasty.
* Agree to join this study and sign the informed consent.

Exclusion Criteria:

* Severe cervical spine kyphosis.
* Cervical spine radiculopathy.
* Laminoplasty with fusion.
* Cervical spine anterior column lesion because of tumor, trauma or infection.
* Severe osteoporosis.
* Morbid obesity.
* patients with mental disorder.
* Pregnancy.
* History of infection within last 3 months.
* Severe nervous system disease.
* Abnormal laboratory report of liver function, kidney function and hematologic system.
* Poor compliance.
* Patients with other surgical contraindications.
* Patients with intemperance or taking drugs.
* Patients who joined other study within the last 3 months.
* Patients with a chief complaint of neck pain (VAS score ≥3 points).
* Left handedness.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with CSM undergoing C3-7 open-door laminoplasty.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram analysis | 3 months after surgery.
  Electroencephalogram analysis (focus on the gamma oscillation at prefrontal cortex) at 3-month follow-up.
Electroencephalogram analysis | 1 year after surgery.
  Electroencephalogram analysis (focus on the gamma oscillation at prefrontal cortex) at 1-year follow-up.
Visual analogue scale for axial pain | 3 months after surgery.
  Visual analogue scale for axial pain before operation and at 3-month follow-up
Visual analogue scale for axial pain | 1 year after surgery.
  Visual analogue scale for axial pain before operation and at 1-year follow-up

SECONDARY OUTCOMES:
Outcome of cervical spine function | 3 months after surgery.
  Neck Disability Index score before operation and at 3-month follow-up
Outcome of cervical spine function | 1 year after surgery.
  Neck Disability Index score before operation and at 1-year follow-up
Quality of life outcome | 3 months after surgery.
  SF-36 score before operation and at 3-month follow-up
Quality of life outcome | 1 year after surgery.
  SF-36 score before operation and at 1-year follow-up
Psychological measures | 3 month after surgery.
  Beck Depression Inventory score before operation and at 3-month follow-up
Psychological measures | 1 year after surgery.
  Beck Depression Inventory score before operation and at 1-year follow-up
Psychological measures | 3 month after surgery.
  Beck Anxiety Inventory score before operation and at 3-month follow-up
Psychological measures | 1 year after surgery.
  Beck Anxiety Inventory score before operation and at 1-year follow-up
Trail Making Test | 3 month after surgery.
  Trail Making Test before operation and at 3-month follow-up
Trail Making Test | 1 year after surgery.
  Trail Making Test before operation and at 1-year follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ming Yi, Beijing, Beijing Municipality
  - Feifei Zhou, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No